CLINICAL TRIAL: NCT02878265
Title: The Effect of Vitamin A With and Without Zinc and Multivitamin Supplementation on Malaria Morbidity in Ghanaian Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Ghana (Other)
Collaborators: Kwame Nkrumah University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wilhelmina Annie Mensah, Ms, University of Ghana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAZ20016
Record Dates: First submitted 2016-08-16; First posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Malaria
Keywords: malaria; vitamin A; Zinc; Multivitamin
MeSH Terms: conditions — Malaria | interventions — Vitamin A; Zinc; Geritol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vitamin A (Placebo Comparator): A single dose of 20,000IU Vitamin A for the whole study period
  Interventions: Dietary Supplement: Vitamin A
- Vitamin A and zinc (Active Comparator): A single dose of 20,000IU Vitamin A and 10mg of elemental zinc each day for 5 months
  Interventions: Dietary Supplement: Vitamin A and ZInc
- Vitamin A , Zinc and Multivitamin (Active Comparator): A single dose of 20,000IU Vitamin A , 10mg of elemental zinc each day and 0.5ml/kg multivitamin syrup for 5 months
  Interventions: Dietary Supplement: Vitamin A , Zinc and Multivitamin

INTERVENTIONS:
Dietary Supplement: Vitamin A — Vitamin A supplements
  Other Names: VA
  Arms: Vitamin A
Dietary Supplement: Vitamin A and ZInc — Combination of vitamin A and zinc supplements
  Other Names: VAZ
  Arms: Vitamin A and zinc
Dietary Supplement: Vitamin A , Zinc and Multivitamin — Combination of vitamin A, zinc and multivitamins
  Other Names: VAZM
  Arms: Vitamin A , Zinc and Multivitamin

SUMMARY:
The aim of this study was to determine the effect of combining vitamin A (VA), zinc (Z) and multivitamins (MV- A, B1, B2, B6, B12, C, D and E) on malaria morbidity

DETAILED DESCRIPTION:
A total of 542 children aged between 6-59 months received either: (i) VA (control) or (ii) VA & Z (VAZ) or (iii) VA, Z & MV (VAZM). VA was delivered as a single dose while MV and Z were delivered daily. Malaria cases were managed by community health workers, who used rapid diagnostic test to confirm infection prior to treatment.

ELIGIBILITY:
Inclusion Criteria:

* under 5years
* will stay in the community for 10years

Exclusion Criteria:

* chronic diseases

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 547 (Actual)
Dates: Start 2011-11; Primary Completion 2012-05 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Incidence of clinical malaria attacks | Baseline and every month up to six months
  While taking the supplement, malaria incidence will be measured

SECONDARY OUTCOMES:
Incidence of diarrhea attacks | Every month up to six months
  While taking the supplement, diarrhea incidence will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Patricia k Brown, PhD, Study Chair — Kwame Nkrumah Univeristy of Science and Technolgy; Wilhelmina A Mensah, Mphil, Principal Investigator — University of Ghana
Locations (1):
- Amoako, Accra, Accra, Ghana

IPD SHARING:
Plan to Share IPD: Yes
To meet the participants and explain the results of their data to them

REFERENCES:
- [Background] Veenemans J, Milligan P, Prentice AM, Schouten LR, Inja N, van der Heijden AC, de Boer LC, Jansen EJ, Koopmans AE, Enthoven WT, Kraaijenhagen RJ, Demir AY, Uges DR, Mbugi EV, Savelkoul HF, Verhoef H. Effect of supplementation with zinc and other micronutrients on malaria in Tanzanian children: a randomised trial. PLoS Med. 2011 Nov;8(11):e1001125. doi: 10.1371/journal.pmed.1001125. Epub 2011 Nov 22. PMID 22131908
- [Result] Zeba AN, Sorgho H, Rouamba N, Zongo I, Rouamba J, Guiguemde RT, Hamer DH, Mokhtar N, Ouedraogo JB. Major reduction of malaria morbidity with combined vitamin A and zinc supplementation in young children in Burkina Faso: a randomized double blind trial. Nutr J. 2008 Jan 31;7:7. doi: 10.1186/1475-2891-7-7. PMID 18237394
- [Result] Owusu-Agyei S, Newton S, Mahama E, Febir LG, Ali M, Adjei K, Tchum K, Alhassan L, Moleah T, Tanumihardjo SA. Impact of vitamin A with zinc supplementation on malaria morbidity in Ghana. Nutr J. 2013 Sep 23;12:131. doi: 10.1186/1475-2891-12-131. PMID 24330422
- [Result] Imdad A, Herzer K, Mayo-Wilson E, Yakoob MY, Bhutta ZA. Vitamin A supplementation for preventing morbidity and mortality in children from 6 months to 5 years of age. Cochrane Database Syst Rev. 2010 Dec 8;(12):CD008524. doi: 10.1002/14651858.CD008524.pub2. PMID 21154399